CLINICAL TRIAL: NCT01913093
Title: N-PhenoGENICS: Neurocognitive-Phenome, Genome, Epigenome and Nutriome In Childhood Leukemia Survivors
Acronym: NPG
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Cancer Society (CCS) (Other); C17 Council (Other); Garron Family Cancer Centre (Other); Pediatric Oncology Group of Ontario (Other)
Responsible Party: Principal Investigator, Shinya Ito, Division Head, Clinical Pharmacology and Toxicology, The Hospital for Sick Children
Other Study IDs: 1000033923
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Childhood Leukemia Survivors
Keywords: Childhood leukemia survivors; Acute lymphoblastic leukemia; Leukemia; Late effects; Folate; Blood folate; Neurotoxicity; Methotrexate; Pharmacogenetics; Cognitive; Cognitive late effects; N-PhenoGENICS
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Neurotoxicity Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA samples obtained via blood, saliva and buccal sample collection.

GROUPS / COHORTS (2):
- Leukemia survivors with neurocognitive deficit: Leukemia survivors with neuro-cognitive deficit phenotype. Based on DIVERGET and other phenotyping tools, we will identify those with the deficit phenotype. This will be treated as "case".
- Leukemia survivors without neurocognitive deficit: Leukemia survivors who did not show impaired neurocognitive function, compared to the Control group defined above.

SUMMARY:
To find possible therapeutic targets to help prevent long-term brain and behavioural side effects in survivors of childhood leukemia that may have been caused by chemotherapy (Treatment-Related late Adverse Neuro-Cognitive Effects: TRANCE). The study hypothesis is that genetic variations of the elements in the folate-related cycles and methotrexate disposition networks are associated with the deficit phenotype (TRANCE) of childhood leukemia survivors.

DETAILED DESCRIPTION:
Hypothesis Genetic variants of the elements in the folate-related cycles and methotrexate disposition networks are associated with the TRANCE phenotype of childhood leukemia survivors.

Objectives

1. To identify TRANCE phenotypes of the childhood leukemia survivors.
2. To characterize the folate and vitamin B12 levels of these children
3. To identify DNA methylation patterns associated with TRANCE trait in the leukemia survivors
4. To identify SNPs associated with the TRANCE trait in the leukemia survivors.
5. To identify the "deficit genotype" associated only with the TRANCE leukemia survivors, but not with general population children who show developmental phenotypes similar to TRANCE: TRANCE-unique deficit variant
6. To replicate the association between the TRANCE-unique deficit variants and the TRANCE trait in a population of childhood leukemia survivors.
7. To evaluate the importance of rare genetic variants in the TRANCE trait in the leukemia survivors.

Study design: A case-control study of leukemia survivors

Analyses

1. Leukemia survivors will be characterized by their status of neurocognitive function, and categorized into the Deficit case and the non-deficit Control case.
2. They will be also characterized by the following attributes

   1. Pathway-based genetic variant status (folate and PK-related genes)
   2. Folate and vitamin B12 status
   3. Epigenetic markers
3. Comparative analyses between neuro-cognitiive deficit phenotype (TRANCE) and Control on those parameters

ELIGIBILITY:
Inclusion Criteria:

* Past diagnosis of acute lymphoblastic leukemia
* 8 years : 0 months - 20 years : 11 months old at the time of their study visit
* At least 2 years : 0 months from the last treatment for acute lymphoblastic leukemia at the time of their study visit
* Continuous complete remission and undergone no bone marrow transplantation or cranial radiation therapy
* Fluent in English (a subject and one parent) for test completion
* Signed informed consent

Exclusion Criteria:

* Inability to complete the phenotyping tests
* Down Syndrome diagnosis

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Childhood leukemia survivors
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
DIVERGET | Within 6 months from the enrolment
  This is a short battery of tests that has been shown to be predictive of both global and academic impairment in survivors of childhood cancer. All neuro-cognitive tests are done on a same day.
Stop Signal Task (SST) | Within 6 months from the enrolment
  Response inhibition, disturbed by behavioral inattention, will be characterized using our task-based computer program, the Stop Signal Task (SST). All neuro-cognitive tests are done on a same day.
CONNERS 3 | Within 6 months from the enrolment
  To characterize behavioural aspects, we will administer the standard measure based on parent report. All neuro-cognitive tests are done on a same day.
Pathway-based gene variant status | Within 3 months from the end of enrolment
  In the hypothesis-driven genome-wide approach, we will focus on the candidate pathways/regions including (but not limited to): a) Folate/methionine cycle genes and transporters; b) drug metabolizing enzymes and transporters (including families of CYP, SLC and ABC transporters); c) epigenetic modifying factors; and d) neuro-regeneration and tissue repair.

SECONDARY OUTCOMES:
WISC-IV | Within 6 months from the enrolment
  In order to confirm validity of DIVERGT in our sample, and provide the data source for future studies, we will include tests of general cognitive function (WISC-IV). All neuro-cognitive tests are done on a same day.
WIAT-III numerical operations and math fluency composite score | Within 6 months from the enrolment
  In order to confirm validity of DIVERGT in our sample, and provide the data source for future studies, we will include tests of general cognitive function: WIAT-III numerical operations and math fluency composite score. All neuro-cognitive tests are done on a same day.
Brief Rating Inventory of Executive Function (BRIEF) | Within 6 months from the enrolment
  In order to confirm validity of DIVERGT in our sample, and provide the data source for future studies, we will administer Brief Rating Inventory of Executive Function (BRIEF), which is designed to assess executive functioning in the home environment. All neuro-cognitive tests are done on a same day.
N-Back Task | Within 6 months from the enrolment
  In order to confirm validity of DIVERGT in our sample, and provide the data source for future studies, we will administer N-Back Task, which is a continuous performance computerized task used to measure aspects of working memory. All neuro-cognitive tests are done on a same day.
Folate, vitamin B12 and iron intake | Within 6 months from the enrolment
  Folate and other vitamin intakes vary among individuals. Folic acid fortification in Canadian food product has changed the Canadian population norm of folate status, virtually eliminating folate deficiency status. However, a large inter-individual variation still remains. We will use a Supplement Questionnaire to capture information on all and any supplements that participants may be currently taking.
Folate status | Within 6 months from the enrolment
  In order to complement the Supplement Questionnaire (above), we will measure the folate concentration in plasma and red blood cells.
Serum vitamin B12 | Within 6 months from the enrolment
  Vitamin B12 and folate pathways interact to maintain biochemical homeostasis. To complement the intake assessment (above), we will measure serum vitamin B12.
Iron status | Within 6 months from the enrolment
  Iron status affects cognitive function of children. In addition to the intake assessment (above), we will estimate iron status by measuring hemoglobin and soluble transferrin receptor.

OTHER OUTCOMES:
Epigenetics marker | Within 3 months from the end of enrolment
  DNA methylation signals represent one of the most stable epigenetic markers, which are known to be affected by environmental factors including drugs and nutrients such as folate. Environmental information conveyed through these factors is translated into gene expression changes mediated by DNA methylation. Although this may contribute to neuro-cognitive deficits of the leukemia survivors, there is no prior data in this regard. Therefore, the aim of this exploratory analysis is to determine if there is any indication that DNA methylation patterns are altered in the participants. DNA will be isolated from each of the blood, buccal swab, and saliva samples and modified using sodium bisulfite, which will then be used to determine DNA methylation patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Shinya Ito, MD, Principal Investigator — The Hospital for Sick Children; Dr. Sharon Guger, Principal Investigator — The Hospital for Sick Children; Dr. Johann Hitzler, Principal Investigator — The Hospital for Sick Children; Dr. Deborah L O'Connor, Principal Investigator — The Hospital for Sick Children; Dr. Russell Schachar, Principal Investigator — The Hospital for Sick Children; Dr. Brenda Spiegler, Principal Investigator — The Hospital for Sick Children; Dr. Rosanna Weksberg, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada